CLINICAL TRIAL: NCT03333772
Title: Feasibility of a Complex Behavioral Intervention for Young Adults With Diabetes: The Resilient, Empowered, Active Living-Telehealth (REAL-T) Study
Brief Title: Feasibility of Delivering a Complex Behavioral Intervention for Young Adults With Diabetes Via Telehealth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Elizabeth Pyatak, Assistant Professor, University of Southern California
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: REAL-T Feasability
Record Dates: First submitted 2017-11-02; First posted 2017-11-07 (Actual); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- REAL-T Intervention (Experimental): The current feasibility study will evaluate the feasibility of implementing the REAL-T RCT by enrolling 10 participants who are 18-30 years of age, conducting the REAL-T intervention with all participants over a 3-month period, evaluating pre-to-post changes in their health and quality of life, and assessing the process of implementing the study (feasibility and participant satisfaction).
  Interventions: Behavioral: REAL-T Intervention

INTERVENTIONS:
Behavioral: REAL-T Intervention — Individualized lifestyle intervention conducted via internet-based videoconferencing and incorporating the following topics: Diabetes knowledge; access to healthcare; communication with healthcare providers; incorporation of diabetes self-care tasks within daily habits and routines; social support; and emotional well-being. Participants will have approximately 6-10 sessions lasting about one hour each, over a 3-month period.

SUMMARY:
Feasibility of a Complex Behavioral Intervention for Young Adults with Diabetes: The Resilient, Empowered, Active Living-Telehealth (REAL-T) Study will evaluate the feasibility of implementing a diabetes management intervention via telehealth in preparation for a large-scale randomized controlled trial (RCT) entitled Evaluation of a Complex Behavioral Intervention for Young Adults with Diabetes: The Resilient, Empowered, Active Living-Telehealth (REAL-T) Study.

DETAILED DESCRIPTION:
Feasibility of a Complex Behavioral Intervention for Young Adults with Diabetes: The Resilient, Empowered, Active Living-Telehealth (REAL-T) feasibility study will evaluate the feasibility of implementing a diabetes management intervention via telehealth in preparation for a large-scale RCT.

Young adulthood is a challenging life stage for many individuals with diabetes; only 17% of YAs age 18-25 and 30% age 26-30 attain recommended A1C targets, and fewer than 1/3 perform self-care in accordance with national guidelines. Yet, it is a crucial stage for establishing health habits that persist throughout adulthood. To address these issues, our research team developed REAL Diabetes (Resilient, Empowered, Active Living with Diabetes), a 6-month individually tailored occupational therapy intervention focused on incorporating diabetes self-care into participants' daily habits and routines, and evaluated its efficacy in a pilot randomized controlled trial (n=81). REAL was shown in intention-to-treat analysis to significantly improve A1C (0.9% reduction; p=0.01) and diabetes-related quality of life (p=0.04). While REAL was highly promising in terms of its positive impact on health and quality of life, the intervention was delivered through home visits, limiting its potential for broad dissemination. Given that our target population experiences significant logistical barriers to clinic attendance (the impetus for our in-home treatment model), we therefore will adapt REAL to be delivered via telehealth (REAL-T), a highly promising care delivery model, and evaluate REAL-T in a large-scale RCT.

The current feasibility study will evaluate the feasibility of implementing the REAL-T intervention via telehealth by enrolling 10 participants who are 18-30 years of age, conducting the REAL-T intervention with all participants over a 3-month period, and assessing the process of implementing the study (feasibility and participant satisfaction).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with either type 1 diabetes or type 2 diabetes for at least 12 months
* Hemoglobin A1C >7.5%
* Resident of Los Angeles County with no imminent plans to relocate
* Fluent in English
* Previous participant in REAL Diabetes Study

Exclusion Criteria:

* Pregnant or planning to become pregnant within the next 4 months
* Diagnosed with a comorbid cognitive or intellectual disability

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2018-02-10 (Actual); Study Completion 2018-02-10 (Actual)

PRIMARY OUTCOMES:
Feasibility | 3 months
  Both formative and summative data will be gathered throughout the study to assess feasibility, defined herein as the extent to which the intervention can be successfully delivered via telehealth. Feasibility will be assessed through surveys.
Acceptability | 3 months
  Both formative and summative data will be gathered throughout the study to assess acceptability, defined herein as the perception of the intervention as agreeable/satisfactory. Acceptability will be assessed through interviews.

SECONDARY OUTCOMES:
Change from baseline in Audit of Diabetes-Dependent Quality of Life (ADD-QoL) at post-intervention | Baseline, 3 months
  19-item survey measure assessing impact of diabetes on social, physical, and emotional functioning
Change from baseline in The Diabetes Empowerment Scale-Short Form (DES-SF) at post-intervention | Baseline, 3 months
  8 item survey measure assessing the psychosocial self-efficacy of people with diabetes
Change from baseline in Problem Areas in Diabetes (PAID) survey at post-intervention | Baseline, 3 months
  5 item survey measure assessing diabetes-related stress
Change from baseline in Patient Health Questionnaire-8 (PHQ-8) survey at post-intervention | Baseline, 3 months
  8-item survey measure assessing severity of depressive symptoms
Change from baseline in Summary of Diabetes Self-Care Activities (SDSCA) at post-intervention | Baseline, 3 months
  14 item survey assessing diet, physical activity, medication adherence and other self-care behaviors relevant to diabetes
Change from baseline in Glycated hemoglobin (HbA1C) at post-intervention | Baseline, 3 months
  Measure of average blood glucose concentration over approximately the previous 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Pyatak, PhD, OTR/L, Principal Investigator — University of Southern California
Locations (1):
- USC Center for Health Professionals, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pyatak EA, Florindez D, Peters AL, Weigensberg MJ. "We are all gonna get diabetic these days": the impact of a living legacy of type 2 diabetes on Hispanic young adults' diabetes care. Diabetes Educ. 2014 Sep-Oct;40(5):648-58. doi: 10.1177/0145721714535994. Epub 2014 May 27. PMID 24867918
- [Background] Pyatak EA, Sequeira PA, Whittemore R, Vigen CP, Peters AL, Weigensberg MJ. Challenges contributing to disrupted transition from paediatric to adult diabetes care in young adults with type 1 diabetes. Diabet Med. 2014 Dec;31(12):1615-24. doi: 10.1111/dme.12485. Epub 2014 May 26. PMID 24798586
- [Background] Pyatak EA, Florindez D, Weigensberg MJ. Adherence decision making in the everyday lives of emerging adults with type 1 diabetes. Patient Prefer Adherence. 2013 Jul 29;7:709-18. doi: 10.2147/PPA.S47577. Print 2013. PMID 23935361
- [Background] Pyatak EA, Carandang K, Davis S. Developing a Manualized Occupational Therapy Diabetes Management Intervention: Resilient, Empowered, Active Living With Diabetes. OTJR (Thorofare N J). 2015 Jul;35(3):187-94. doi: 10.1177/1539449215584310. PMID 26594741
- [Background] Pyatak EA, Carandang K, Vigen C, Blanchard J, Sequeira PA, Wood JR, Spruijt-Metz D, Whittemore R, Peters AL. Resilient, Empowered, Active Living with Diabetes (REAL Diabetes) study: Methodology and baseline characteristics of a randomized controlled trial evaluating an occupation-based diabetes management intervention for young adults. Contemp Clin Trials. 2017 Mar;54:8-17. doi: 10.1016/j.cct.2016.12.025. Epub 2017 Jan 5. PMID 28064028